CLINICAL TRIAL: NCT06334146
Title: Feasibility and Acceptability of Tap Dance as a Therapeutic Intervention for Adults With Lower Limb Amputation
Brief Title: Tap Dance for Adults With Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Jenny Kent, Assistant Professor, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2023-62
Record Dates: First submitted 2024-02-26; First posted 2024-03-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Amputation; Traumatic, Leg, Lower

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tap dance program (Experimental): Participants undertake tap dance program.
  Interventions: Other: Tap dance program

INTERVENTIONS:
Other: Tap dance program — Participants will take part in a weekly adapted tap dance class, for one hour per week, for eight weeks.

SUMMARY:
The goal of this study is to determine whether it is possible for people with lower limb amputation (LLA) to perform adapted tap dance, whether an adapted tap dance program would be enjoyable, and whether it may improve balance and balance confidence.

There is a lack of research investigating therapeutic interventions for people with lower limb amputation (LLA). Tap dance encourages balance and novel movements of the limbs, while providing auditory feedback from the feet that provide information about the foot's contact with the ground, which may help prosthesis users gain a better ability to understand where their prosthetic foot is in space. As with most forms of dance, tap is usually taught and practiced in a group setting, which encourages community involvement. It has been shown to be safer than many forms of dance due to low impact forces. It also, as a genre, can incorporate canes, chairs and partner work, providing the ability to modify steps/moves when required so that they remain practical, achievable and safe for people with mobility limitations, while still enabling participation. It therefore may be an accessible dance medium to help improve balance, balance confidence, and build community for people with LLA.

Participants will be asked to:

* come to 1 hour dance classes, once per week, for 8 weeks.
* do mobility tests before and after the program
* complete questionnaires before, during and after the program. The total time for participation is approximately 8-10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral lower limb amputation at ankle level or above
* fitted with a walking prosthesis, used regularly for walking in the home and the community
* good socket fit
* able to stand or walk for 2 minutes at a time with or without an assistive device
* willing to travel to the University of Nevada Las Vegas for tap classes once a week for 8 weeks, and for two testing sessions
* able to complete all required outcome measures
* able to understand written and spoken English

Exclusion Criteria:

* leg/foot ulcer/sore or other conditions that cause pain during weight-bearing
* cardiovascular, respiratory or other critical health conditions that preclude moderate physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Session Adherence | through study completion, over 8 weeks
  Number of planned dance tap sessions attended
Physical Activities Enjoyment Scale (PACES) | Intervention week 8
  Total score on 18-item self response scale measuring enjoyment of an activity, out of a maximum 126.

SECONDARY OUTCOMES:
Change in Timed Up-and-Go test score | 8 weeks
  Timed walking test in which the participant rises from a chair, walks to a marker 10 feet away, turns, and returns to sit in the chair. Time to complete, in seconds, is recorded.
Change in Four Square Step Test score | 8 weeks
  Time taken in seconds to complete a stepping sequence between two canes placed in a cross shape.
Change in Berg Balance Scale score | 8 weeks
  Score out of 23, for performance of 14 mobility-related tasks.
Change in Activities-Specific Balance Confidence Scale score | 8 weeks
  16 item self response scale measuring balance confidence. Scored out of 100%
Physical Activities Enjoyment Scale (PACES) score - Mid program | Intervention week 4
  Total score on 18-item self response scale measuring enjoyment of an activity, out of a maximum 126.
Change in Trinity Amputation and Prosthesis Experience Scale (TAPES) functional activity restriction subscale score | 8 weeks
  Total score on functional activity restriction subscale of the TAPES - self reported outcome measure, out of maximum 12
Change in Trinity Amputation and Prosthesis Experience Scale (TAPES) social activity restriction subscale score | 8 weeks
  Total score on social activity restriction subscale of the TAPES - self reported outcome measure, out of maximum 12
Change in Trinity Amputation and Prosthesis Experience Scale (TAPES) athletic activity restriction score | 8 weeks
  Total score on athletic activity restriction subscale of the TAPES - self reported outcome measure, out of maximum 12
Use of assistive devices per session | through study completion, over 8 weeks
  Percentage of sessions for which assistive devices are used
Session completion per session | through study completion, over 8 weeks
  Percentage of planned dance tap sessions completed

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Kent, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No